CLINICAL TRIAL: NCT05515016
Title: A Fatty Flap Sculpted From the Double Chin for a Better Face Profile: an Original Technique
Brief Title: A Fatty Flap Taken From the Double Chin for Chin Enhancement: a New Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Tahar Maamouri University Hospital (Other)
Responsible Party: Principal Investigator, Imen Turki Mehri, MD, Principal investigator, Mohamed Tahar Maamouri University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Maamouri Teaching hospital
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Adiposity; Micrognathism
Keywords: Retrognathia; Mandibular advancement; Adipose tissue; Cervicoplasty
MeSH Terms: conditions — Obesity; Micrognathism; Retrognathia

STUDY DESIGN:
Intervention Model Description: The same surgical procedure was performed on 10 participants. These participants had a double chin with skin redundancy and a receding chin. The result was evaluated with photos and chin advancement was measured with a Vernier caliper.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A surgical technique for double chin treatment and chin advancement (Other): the same surgical technique was performed on 10 participants with their consent. Subplatysmal fat, of the submental region, was dissected from the subcutaneous plan and the platysma muscle, then elevated as a flap to be plicated and turned, then fixed on the muscular layer of the chin. This technique provides both double chin treatment and chin advancement. It improves the profile of the face.
  Interventions: Procedure: chin enhancement with a fatty flap sculpted from the double chin

INTERVENTIONS:
Procedure: chin enhancement with a fatty flap sculpted from the double chin — Under general anesthesia, an incision was made behind the submental crease followed by the excision of the skin excess. The preplatysmal fatty compartment was individualized through a subcutaneous dissection. Then, the lower part of the preplatysmal fat was cut to start its separation from the platysma muscle, thus obtaining a real vascularized fatty flap. This flap could be folded on itself, then easily turned over to be fixed on the muscular layer of the chin.
  Other Names: submental fatty flap treating the double chin and correcting the micrognathia

SUMMARY:
The double chin is a troublesome component of the lower third of the face. It gives an embarrassing and unpleasant facial appearance to both men and women leading them to ask for liposuction. Moreover, a "receding chin" causes blunting of the cervico-mental angle, a fleshy appearing neck, a disproportion in the profile line of the face with a prominent looking nose, and an irregular mandibular border. This study is about an innovative surgical procedure: Instead of doing liposuction of the double chin, the investigators used the fat of this area as a flap to improve a "receding chin". hence both the double chin and the receding chin are treated.

DETAILED DESCRIPTION:
the surgical technique was performed on 10 participants. written informed consent was obtained from all the participants.

Description of the surgical technique:

The investigators began by delineating the undesirable subplatysmal fat located in the submental region, just below the subcutaneous fat. The skin redundancy assessed by the pinch test was excised. Under general anesthesia, an incision was made behind the submental crease followed by the excision of the skin excess. The subplatysmal fatty compartment was individualized through a subcutaneous dissection. Then, the lower part of the subplatysmal fat was cut to start its separation from the platysma muscle, thus obtaining a real vascularized fatty flap. This flap could be folded on itself, then easily turned over to be fixed on the thin layer of the pre-muscular fat overlying the chin. Hemostasis was performed correctly avoiding the establishment of drainage.

chin projection and submental rejuvenation were obtained. The advancement of the chin ranged from 3,5 to 12 millimeters. The stability of the translated fat was observed after surgery for more than two years.

ELIGIBILITY:
Inclusion Criteria:

* the presence of a "double chin" with slightly redundant skin and a "receding chin" causing a fleshy appearing neck, and a disproportion in the face profile

Exclusion Criteria:

* any history of a precedent surgery on the neck, the presence of a traumatic or a burn scar on the cervical region.

Ages: 45 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Chin advancement measure | The change of chin projection at 6 months after the surgical procedure
  For the objective evaluation: Chin advancement was evaluated by measuring, with a Vernier caliper, the distance between the submental crease and the soft tissue at the pogonion. This distance was taken before and after the surgical procedure. The advancement of the chin ranged from 3,5 to 12 millimeters (mm). This measurement was taken by the investigator during the follow-up appointments. For the subjective evaluation: The results were evaluated on patient reviews and photographic studies (before and after surgery).
Chin advancement measure | The change of chin projection at 12 months after the surgical procedure
  For the objective evaluation: Chin advancement was evaluated by measuring, with a Vernier caliper, the distance between the submental crease and the soft tissue at the pogonion. This distance was taken before and after the surgical procedure. The advancement of the chin ranged from 3,5 to 12 millimeters (mm). This measurement was taken by the investigator during the follow-up appointments. For the subjective evaluation: The results were evaluated on patient reviews and photographic studies (before and after surgery).
Chin advancement measure assessing the stability of the result | The change of chin projection at 24 months after the surgical procedure
  For the objective evaluation: Chin advancement was evaluated by measuring, with a Vernier caliper, the distance between the submental crease and the soft tissue at the pogonion. This distance was taken before and after the surgical procedure. The advancement of the chin ranged from 3,5 to 12 millimeters (mm). This measurement was taken by the investigator during the follow-up appointments. For the subjective evaluation: The results were evaluated on patient reviews and photographic studies (before and after surgery).
Fat deposits removal in the submental region | At 6 months after the surgical procedure
  This outcome was evaluated on photos (face and profile) before and after surgery. A questionnaire including three levels of satisfaction (not satisfied, satisfied, very satisfied) was completed by the participants concerning the surgical outcomes including the submental change and the chin advancement.
Fat deposits removal in the submental region | At 12 months after the surgical procedure
  This outcome was evaluated on photos (face and profile) before and after surgery. A questionnaire including three levels of satisfaction (not satisfied, satisfied, very satisfied) was completed by the participants concerning the surgical outcomes including the submental change and the chin advancement.

SECONDARY OUTCOMES:
The evaluation of the surgical scar | At 6 months after the surgical procedure
  The aspect of the scar was evaluated by the investigator by two parameters: the pigmentation (normal colored, hypopigmentation, hyperpigmentation) and the throphycity (hypertrophic, depressive, adequate trophicity).
The evaluation of the surgical scar | At 12 months after the surgical procedure
  The aspect of the scar was evaluated by the investigator by two parameters: the pigmentation (normal colored, hypopigmentation, hyperpigmentation) and the throphycity (hypertrophic, depressive, adequate trophicity).

CONTACTS AND LOCATIONS:
Overall Officials: IMEN T MEHRI TURKI, Dr, Principal Investigator — Teaching hospital Mohamed Tahar Maamouri, nabeul

REFERENCES:
- [Result] Shamban AT. Noninvasive Submental Fat Compartment Treatment. Plast Reconstr Surg Glob Open. 2016 Dec 14;4(12 Suppl Anatomy and Safety in Cosmetic Medicine: Cosmetic Bootcamp):e1155. doi: 10.1097/GOX.0000000000001155. eCollection 2016 Dec. PMID 28018773
- [Result] Strauss RA, Abubaker AO. Genioplasty: a case for advancement osteotomy. J Oral Maxillofac Surg. 2000 Jul;58(7):783-7. doi: 10.1053/joms.2000.7266. PMID 10883694
- See also: Noninvasive Submental Fat Compartment Treatment — https://pubmed.ncbi.nlm.nih.gov/28018773/
- See also: Genioplasty: a case for advancement osteotomy — https://pubmed.ncbi.nlm.nih.gov/10883694/